CLINICAL TRIAL: NCT00594035
Title: A Prospective, Multi-Center, Randomized Controlled Study to Compare the Spinal Sealant System as an Adjunct to Sutured Dural Repair With Standard of Care Methods During Spinal Surgery
Brief Title: Study to Evaluate Safety and Effectiveness of Spinal Sealant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRS-05-001
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Spinal Procedure Requiring Dura Incision
Keywords: Spinal procedure; Dura incision

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Spinal Sealant
  Interventions: Device: Spinal Sealant System
- 2 (Active Comparator): Standard of care
  Interventions: Device: Standard of care

INTERVENTIONS:
Device: Spinal Sealant System
  Arms: 1
Device: Standard of care — Standard of care: devices intended to provide a watertight closure
  Other Names: (i.e. devices intended to provide a watertight closure)
  Arms: 2

SUMMARY:
To evaluate the safety and efficacy of the Spinal Sealant as an adjunct to sutured dural repair compared with standard of care methods (control) to obtain watertight dural closure in patients undergoing spinal surgery.

DETAILED DESCRIPTION:
Neurosurgical procedures in the spine often involve incision of the dura mater to access the spinal cord. If the dural incision is not properly repaired and watertight closure is not achieved cerebrospinal fluid (CSF) can escape presenting a risk for significant morbidity. The most frequent complication of CSF leak is recurring headache complicated with symptoms of nausea and vomiting. Furthermore fluid collection under skin prevents proper wound healing and may lead to wound breakdown and infection of the incision or both. Persistent CSF leak has also been associated with the development of cerebellar hemorrhage and subdural hematoma. Primary repair and watertight closure are paramount to minimizing risk and sequelae associated with CSF leak.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for an elective spinal procedure that requires a dural incision will be considered for study participation.
* Patient requires a procedure that involving surgical wound classification Class 1/Clean (per CDC criteria)
* Presence of a non-watertight dural closure, either spontaneously or upon Valsala maneuver at 20-25 cm H20 for 5-10 seconds.

Exclusion Criteria:

* Active spinal and/or systemic infection
* Patient requires additional spinal surgery within the study time period
* Patient has had a previous spinal surgery involving dural exposure and/or entry at the same level(s) as the study procedure
* Patient has a pre-existing external lumbar CSF drain or internal CSF shunt
* Patient is participating in a clinical trial of another investigational device or drug
* Patient with creatinine > 2.0 mg/dL
* Patient with total bilirubin > 2.5 mg/dL
* Pregnant or breast-feeding females or females who wish to become pregnant during the length of study participation
* Patient has been treated with chronic steroid therapy (>4 weeks) unless discontinued more than 6 weeks prior to surgery
* Patient has documented history or significant coagulopathy with a PTT >35 sec, PT/INR >1.2, receiving asprin, or NSAIDS at the time of surgery
* Patient receiving warfarin or heparin at the time of surgery
* Patient has a diagnosed and documented compromised immune system and/or autoimmune disease
* Patient has has chemotherapy treatment within 6 months prior to, or planned during the study
* Patient has had prior radiation treatment to the surgical site or has planned radiation therapy within 30 days post procedure
* Patient has known malignancy or other condition with prognosis shorter than 6 months
* Patients with documented history of uncontrolled diabetes
* Patient requires use of synthetic or non-autologous duraplasty material
* Patient has a gap greater than 2mm remaining after primary dural closure
* Patient has undergone laminoplasty decompression
* Patient has undergone a syringomyelia procedure where the shunt is not placed in the subarachnoid position
* Patient has undergone a Chiari Malformation procedure that does not entail a dural incision at or below the C1 level
* The investigator determines that participation in the study may jeopardize the safety or welfare of the patient
* The investigator determines that the patient should not be included in the study for reason(s) not already specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Scerbin, Study Director — Medtronic - MITG
Locations (1):
- Confluent Surgical, Inc., Bedford, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects scheduled for spinal procedures requiring a dural incision were considered for study participation. The Study involved 24 investigational sites within the United States. Subjects were recruited from neurosurgery practices between the period of 01 September 2005 (first subject consented) to 06 Feb 2008 (last visit date).
Pre-assignment Details: Enrollment was considered the point of randomization. Subjects were randomized intra-operatively after confirmation that all pre-operative and intra-operative eligibility criteria had been met.
Groups:
- Spinal Sealant: Subjects that recieve DuraSeal Spinal Sealant
- Standard of Care: Subjects who receive standard or care meathods of dural sealing
Period: Overall Study
Arm/Group | Spinal Sealant | Standard of Care
Started | 102 (102 subjects were randomized to Spinal Sealant) | 56 (56 subjects were randomized to the control group (standard of care))
Completed | 100 (100 Spinal Sealant subjects were evaluable at the 90-day visit) | 53 (53 control group subjects were evaluable at the 90-day visit)
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject transferred to nursing home | 0 | 1
Not completed — Subject couldn't return due to job | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Sealant | Standard of Care | Total
Number analyzed (Participants) | 102 | 56 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 52 | 141
  >=65 years | 13 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.6) | 42.3 (14.5) | 45.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 30 | 84
  Male | 48 | 26 | 74
Region of Enrollment [Number; unit: participants]
  United States | 102 | 56 | 158

OUTCOME MEASURES:

1. Primary Outcome: Watertight Dural Closure
Description: Number of subjects displaying a watertight dural closure after assigned treatment intra-operatively.
Time Frame: Intra-Operative
Measure: Number; unit: Participants
Arm/Group | Spinal Sealant | Standard of Care
Number analyzed (Participants) | 102 | 56
Participants | 102 | 36

ADVERSE EVENTS:
Time Frame: Subjects were followed and adverse events were collected for 90 days after surgery.
Arm/Group | Spinal Sealant | Standard of Care
Serious Adverse Events (participants affected / at risk) | 30/102 | 10/56
Other Adverse Events (participants affected / at risk) | 65/102 | 41/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Sealant (N=102) | Standard of Care (N=56)
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrospinal Fistula (Nervous system disorders) | 2 (2) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Graft Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Incision Site Complication (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Loss of Proprioception (Nervous system disorders) | 1 (1) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sensory Loss (Nervous system disorders) | 1 (1) | 1 (1)
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope Vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Sealant (N=102) | Standard of Care (N=56)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Body Temperature Increased (Investigations) | 46 (48) | 20 (23)
Constipation (Gastrointestinal disorders) | 9 (9) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 12 (16) | 7 (8)
Hyporeflexia (Nervous system disorders) | 7 (7) | 1 (1)
Incision Site Complication (Injury, poisoning and procedural complications) | 12 (14) | 2 (4)
Incision Site Infection (Infections and infestations) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Neuralgia (Nervous system disorders) | 5 (5) | 0 (0)
Pain In extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Paraesthesia (Nervous system disorders) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 19 (23) | 13 (14)
Urinary Retention (Renal and urinary disorders) | 11 (13) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 11 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The sponsor can review results at least 30 days prior to public release, and at the request of Sponsor, the PI will withhold submission for an additional period, not to exceed 90 days.
* The first publication of the study results shall be made in conjunction with a joint, multi-center publication of the results. If a multi-center publication is not submitted within 12 months after the conclusion of the Study, the PIs may publish the results from their individual site.